CLINICAL TRIAL: NCT06613633
Title: Pattern of Failure and Feasibility of Consolidative Stereotactic Radiotherapy in Third-generation EGFR-TKI-treated Metastatic EGFR-mutant Non-small Cell Lung Cancer: A Prospective, Observational Study
Brief Title: Third-generation EGFR-TKI Treatment in Metastatic EGFR-mutant NSCLC
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Collaborators: Shanghai Chest Hospital (Other); Wuhan TongJi Hospital (Other)
Responsible Party: Principal Investigator, Zhengfei Zhu, Professor, Fudan University
Other Study IDs: 2018-NSCLCSIB
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-10

CONDITIONS: Third-generation TKI; NSCLC (Advanced Non-small Cell Lung Cancer)
Keywords: NSCLC; EGFR
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; aumolertinib; aflutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- third-generation EGFR-TKI monotherapy
  Interventions: Drug: third-generation EGFR-TKI (Osimertinib, Almonertinib or Furmonertinib)

INTERVENTIONS:
Drug: third-generation EGFR-TKI (Osimertinib, Almonertinib or Furmonertinib) — Patients with advanced EGFR-mutated NSCLC who met the inclusion criteria and received third-generation EGFR-TKI (monotherapy or combined with brain radiotherapy)

SUMMARY:
The goal of this observational study is to explore the feasibility of stereotactic radiotherapy (SRT) as consolidation therapy for patients with advanced non-small-cell lung cancer who were treated with third-generation epidermal growth factor receptor-tyrosine kinase inhibitor (EGFR-TKI). The investigators plan to explore the time to achieve the best response after EGFR-TKI treatment, the characteristics of the distribution of lesions when the best response is achieved, the feasibility of SRT when the best response is achieved, and the phenotype of disease progression after EGFR-TKI resistance.

In summary, this study will provide critical information for exploring the feasibility and optimal design of SRT as consolidation therapy for advanced NSCLC patients treated with third-generation EGFR-TKI, which will further promote the optimization of comprehensive treatment for EGFR-mutant advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed non-small cell lung cancer;
* clinical stage IV (AJCC, 8th edition, 2017);
* EGFR sensitizing mutations (L858R or 19del);
* age≥18 years old;
* KPS score≥70;
* complete systemic imaging (including brain MRI) before third-generation EGFR-TKI treatment;
* received standard third-generation EGFR-TKI therapy (monotherapy or combined with brain radiotherapy);
* willing to cooperate with the follow-up after third-generation EGFR-TKI treatment;
* informed consent of the patient.

Exclusion Criteria:

* Multiple primary or metastatic tumors (except early skin cancer, cervical carcinoma in situ that has been treated radically, with no recurrence or progression for more than 5 years);
* Pregnant or lactating women who, as judged by the investigator, were not candidates for brain MRI;
* Uncontrolled epilepsy, central nervous system disease, or history of mental disorders, judged by the researcher to potentially interfere with the signing of the informed consent form or affect patient compliance.;
* patients without EGFR sensitive mutations or with unknown EGFR mutation status.

Withdrawal criteria

* The investigators considered that the patients had poor adherence to the study protocol.
* The patient withdrew informed consent and asked to withdraw.
* There was any safety reason (adverse event) considered by the investigator;
* Due to other underlying diseases, side effects, economic factors, and other reasons, patients did not receive regular doses of third-generation EGFR-TKI (continuous withdrawal time more than 1 week, cumulative withdrawal time more than 2 weeks, etc.).
* The patient was not followed up according to the protocol.
* Other circumstances in which withdrawal from the study was deemed necessary by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced EGFR-mutant NSCLC patients receiving third-generation EGFR-TKIs are enrolled
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-20 (Actual)

PRIMARY OUTCOMES:
Time to Best Response | 5 years
  The time from the first day of third-generation EGFR-TKI treatment to the point at which the smallest tumor burden is observed on imaging studies.

SECONDARY OUTCOMES:
Distribution of Tumor Lesions at Best Response | 5 years
  the distribution of tumor lesions at the time when the smallest tumor burden is observed on imaging. Focus on whether the remaining lesions are suitable for consolidative stereotactic radiotherapy, per the relevant criteria endorsed by the NRG-BR001 study.
Phenotypes of Disease Progression After Third-Generation EGFR-TKI Resistance | 5 years
  Tumor distribution when disease progression occurs during third-generation EGFR-TKI treatment (disease progression is defined by RECIST 1.1 criteria). The pattern of progressive disease will be classified into the following three types based on imaging assessment:
  1. Original Site Failure (OF): Progression of lesions that were present at baseline (enlargement of existing lesions).
  2. Distant Site Failure (DF): New tumor lesions occurring in areas where no lesions were present at baseline.
  3. Original and Distant site failure (ODF): The coexistence of the two situations mentioned above.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality